CLINICAL TRIAL: NCT03769818
Title: Role of Adjuvant Dexamethasone for Erector Spinae Plane Block for Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy: A Randomized, Double-blind Controlled Trial
Brief Title: Role of Dexamethasone for Erector Spinae Plane Block in Patients Undergoing Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/181/18
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
Keywords: erector spinae plane block; total abdominal hysterectomy; dexamethasone
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: A prospective Randomized Interventional double-blind study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participating patients, surgeons, anesthesiologists and medical investigators who will be involved in the data collection will be all blinded to the patient's group assignment until the collection of data for all cases will be complete for group 1 and 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bupivacaine and dexamethasone (Active Comparator): Bilateral ESP block with 20 ml of 0.25% bupivacaine + 4 mg/kg dexamethasone diluted with isotonic saline.
  Interventions: Drug: bupivacaine; Drug: dexamethasone
- bupivacaine and placebo to dexamethasone (Active Comparator): Bilateral ESP block with 20 ml of 0.25% bupivacaine bilaterally plus placebo to dexamethasone
  Interventions: Drug: bupivacaine; Drug: placebo to dexamethasone
- control group (Placebo Comparator): Bilateral ESP block with placebo to bupivacaine bilaterally plus placebo to dexamethasone
  Interventions: Drug: placebo to dexamethasone; Drug: placebo to bupivacaine

INTERVENTIONS:
Drug: bupivacaine — Bilateral TAP block with 20 ml of 0.25% bupivacaine
  Other Names: Active Comparator
  Arms: bupivacaine and dexamethasone; bupivacaine and placebo to dexamethasone
Drug: dexamethasone — Bilateral TAP block with 4 mg/kg dexamethasone diluted with isotonic saline.
  Other Names: active comparator
  Arms: bupivacaine and dexamethasone
Drug: placebo to dexamethasone — Bilateral TAP block with placebo to dexamethasone.
  Arms: bupivacaine and placebo to dexamethasone; control group
Drug: placebo to bupivacaine — Bilateral TAP block with placebo to bupivacaine.
  Arms: control group

SUMMARY:
The aim to study the efficacy of bupivacaine 0.25% with dexamethasone and that of bupivacaine 0.25% alone for erector spinae plane block for postoperative analgesia in patients undergoing total abdominal hysterectomy Group 1: bupivacaine 0.25% + dexamethasone 8 mg

* Group 2: bupivacaine 0.25%
* Group3: control group A prospective Randomized Interventional double-blind study.

DETAILED DESCRIPTION:
Optimal dynamic analgesia is recognized as the key to enhanced recovery following open abdominal surgery. In the last decade, there has been a significant shift away from thoracic epidural analgesia (TEA) that has been long considered as the gold standard. Various techniques have tried to replicate the analgesic efficacy of TEA. They include transversus abdominis plane analgesia (TAP), rectus sheath analgesia (RS), wound infusion analgesia (WI) and trans muscular quadratus lumborum analgesia. However, each of these techniques has specific limitations that prevent them from being the analgesic technique of choice for all open abdominal surgeries. Chin et al first described the erector spinae plane (ESP) block for providing analgesia following ventral hernia repair. The unique feature of the ultrasound-guided truncal blocks is that in all of these techniques, in contrast to peripheral nerve blocks, no nerve or plexus needs to be identified: Local anesthesia (LA) is injected in a particular muscle plane, in which the injectate spreads and reaches the intended nerves. This simple mechanism has made delivery of nerve blocks easy and versatile.

ELIGIBILITY:
Inclusion Criteria:

* Women ranging age between 30-60 years a who undergoing elective total abdominal hysterectomy

Exclusion Criteria:

* Participants had known sensitivity to bupivacaine
* Participants had difficulty in intubation
* Participants were on chronic pain medication or already on long-term opioids
* Participants smokers
* Participants with disabilities who were unable to communicate pain levels
* refuse to consent

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — patients undergoing total abdominal hysterectomy
Enrollment: 150 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Visual analog score for pain during movement | 24 hours post operative
  movement-evoked pain measurements ranging from 0 to 10, where 0 no pain and 10 maximum pain

SECONDARY OUTCOMES:
Visual analog score for pain during rest | 24 hours postoperative
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
number of patients need Fentanyl consumption | 24 hours postoperative
  calculation of the number of patients need Fentanyl consumption
number of days patients stay in hospital | 4 weeks
  calculation of number of days patients stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided